CLINICAL TRIAL: NCT06058468
Title: Cardioneuroablation of Right Anterior Ganglionated Plexus vs Pulmonary Vein Isolation in Patients With Paroxysmal Atrial Fibrillation and Enhanced Vagal Tone
Brief Title: Cardioneuroablation vs Pulmonary Vein Isolation in Treatment of Paroxysmal Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Centre, Poland (Other)
Responsible Party: Principal Investigator, Piotr Futyma, Professor, St. Joseph's Centre, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/084/W
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Atrial Fibrillation; Vagally-mediated; Cardioneuroablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioneuroablation of right anterior ganglionated plexus (Experimental)
  Interventions: Procedure: Cardioneuroablation of right anterior ganglionated plexus
- Pulmonary vein isolation (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Cardioneuroablation of right anterior ganglionated plexus — Right anterior ganglionated plexus will be localized using anatomical approach. Radiofrequency energy will be delivered until heart rate acceleration >30% is achieved or if radiofrequency time exceeds 120 seconds.
  Arms: Cardioneuroablation of right anterior ganglionated plexus
Procedure: Pulmonary vein isolation — Application sites near the ostia of pulmonary veins will be determined. Radiofrequency energy will be delivered using point-by-point technique. After applications, the acute PVI endpoint will be confirmed by the elimination of PV potentials and lack of capture during pacing from the ablation lines.
  Arms: Pulmonary vein isolation

SUMMARY:
The goal of this study is to compare effectiveness of cardioneuroablation of right anterior ganglionated plexus and pulmonary vein isolation in patients with enhanced vagal tone expressed as deceleration capacity >7.5ms.

DETAILED DESCRIPTION:
Patients included into the study will be randomized to a group undergoing cardioneuroablation (CNA) of the right anterior ganglionated plexus (RAGP) or pulmonary vein isolation (PVI).

In CNA group the location of RAGP will be determined anatomically below the superior vena cava ostium near the superior-septal aspect of the right atrium. Radiofrequency (RF) applications will be delivered and will be continued until heart rate (HR) acceleration >30% is achieved or if the RF time exceeds 120s.

In the PVI group point-by-point RF isolation of all pulmonary veins will be performed.

Clinical follow-up (FU) will consist of multiple ambulatory visits combined with standard ECG readings and a 7-day Holter recording. During FU visits, a detailed history of any palpitations, episodes of atrial fibrillation (AF), and hospitalizations for cardiac arrhythmias will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation documented in ECG or Holter monitoring
* Deceleration capacity >7.5ms
* Life expectancy more than 1 year
* Age ≥18 years

Exclusion Criteria:

* Permanent AF lasting more than one year or persistent AF lasting more than 7 days
* AF secondary to electrolyte imbalance, thyroid disease, alcohol abuse, or other non-heart related causes
* Anteroposterior dimension of the left atrium in the echocardiography ≥43mm
* Clinically significant arrhythmias other than AF
* Significant valvular disease
* Valve prosthesis
* Heart failure III or IV Class in New York Heart Association Classification
* Previous ablation of atrial fibrillation or atrial flutter
* History of a patent foramen ovale/atrial septal defect closure
* History of left atrial appendage closure
* Atrial myxoma
* Presence of a cardiac pacemaker, defibrillator or cardiac resynchronization therapy device
* History of pericarditis
* Congenital heart disease
* History of bleeding or coagulation disorders
* Contraindications to oral anticoagulation
* Contraindications to computed tomography or magnetic resonance imaging
* Pregnancy or breast-feeding
* BMI>31
* History of transplantation
* Severe lung disease
* Chronic renal failure defined as estimated glomerular filtration rate (eGFR) <30 mL/min/m2
* Cancer
* Significant infection
* Life expectancy less than one year
* Mental disorders
* Lack of informed consent to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | 1 year
  AF episode lasting 30 seconds or more, documented on 12-lead ECG, event or Holter monitoring

IPD SHARING:
Plan to Share IPD: No